CLINICAL TRIAL: NCT04195282
Title: Therapeutic Effects and Safety of RL-1 Novel Human-derived Bio-artificial Liver Treatment in Patients of Hepatitis b Virus Related Acute-on-chronic Liver Failure
Brief Title: RL-1 Novel Human-derived Bio-artificial Liver Treatment in Patients of HBV Related ACLF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professer, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PL9
Record Dates: First submitted 2019-12-08; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis B; Acute-On-Chronic Liver Failure
Keywords: hepatitis b virus; acute-on-chronic liver failure; artificial liver
MeSH Terms: conditions — Hepatitis B; Acute-On-Chronic Liver Failure | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma exchange group (Active Comparator): 10 patients will receive conventional treatment plus plasma exchange
  Interventions: Other: Plasma exchange
- RL-1 Novel Human-derived Bio-artificial Liver treatment group (Experimental): 10 patients will receive conventional treatment plus RL-1 Novel Human-derived Bio-artificial Liver treatment
  Interventions: Other: RL-1 Novel Human-derived Bio-artificial Liver Treatment

INTERVENTIONS:
Other: Plasma exchange — Patients will receive treatment of plasma exchange for three times in two weeks. The volume of fresh frozen plasma used in plasma exchange is about 2000 millilitre per time.
  Arms: Plasma exchange group
Other: RL-1 Novel Human-derived Bio-artificial Liver Treatment — Patients will receive RL-1 Novel Human-derived Bio-artificial Liver treatment for three times in two weeks. The volume of plasma exchanged in the system is about 4000 millilitre per time.
  Arms: RL-1 Novel Human-derived Bio-artificial Liver treatment group

SUMMARY:
This study is to investigate the clinical efficacy and safety of RL-1 Novel Human-derived Bio-artificial Liver treatment in patients with Hepatitis b virus related acute-on-chronic liver failure.

DETAILED DESCRIPTION:
Hepatitis b virus (HBV) related acute-on-chronic liver failure (ACLF) is a serious condition with high mortality rate in China. But there still lacks of effective therapies in treatment of HBV related ACLF, except liver transplantation. RL-1 Novel Human-derived Bio-artificial Liver treatment may be an effective and safe therapy due to the previous clinical data. This study is to investigate the clinical efficacy and safety of RL-1 Novel Human-derived Bio-artificial Liver treatment in patients with HBV related ACLF.

ELIGIBILITY:
Inclusion Criteria:

1. Positive hepatitis b surface antigen or hepatitis b virus DNA > 0.5 year;
2. Age from 18 to 65 years old;
3. Serum total bilirubin level > 10 times upper limit of normal;
4. Prothrombin time activity < 40% and ≥30%；
5. Platelets > 50*10 E9/L.

Exclusion Criteria:

1. Other active liver diseases;
2. Hepatocellular carcinoma or other malignancy;
3. Pregnancy or lactation;
4. Human immunodeficiency virus infection or congenital immune deficiency diseases;
5. Severe diabetes, autoimmune diseases;
6. Other important organ dysfunctions;
7. Severe complications including severe infection, gastrointestinal bleeding, hepatic encephalopathy, hepatorenal syndrome;
8. Patients can not follow-up;
9. Investigator considering inappropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 4 week
  All adverse events (i.e. fever, allergy, bleeding, hypotension, thrombosis) are observed in the follow-up.

SECONDARY OUTCOMES:
Survival rate | 4 week
  Whether patients will survive after treatment is observed in the follow-up.
Symptoms | 4 week
  All symptoms (i.e. fatigue, appetite, nausea, vomiting, jaundice, consciousness) are observed in the follow-up.
Blood cells | 4 week
  Blood cells are observed in the follow-up.
Alanine transaminase | 4 week
  Alanine transaminase is observed in the follow-up.
Total bilirubin | 4 week
  Total bilirubin is observed in the follow-up.
Serum creatinine | 4 week
  is observed in the follow-up.
Prothrombin time | 4 week
  Prothrombin time is observed in the follow-up.
Blood ammonia | 4 week
  Blood ammonia is observed in the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China